CLINICAL TRIAL: NCT00378885
Title: The Effect of a Theory Based Tailored Intervention Online on the Reduction of Risk Behavior for HIV Transmission Among Men Who Have Sex With Men - a Randomized, Single-Blind, Active (Waiting-List) Controlled Trial
Brief Title: Effect Study of a Theory-Based Internet Intervention on Safe-Sex Practices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Service of Amsterdam (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: GGD 4013
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2006-09-21 (Estimated); Status verified 2006-09

CONDITIONS: Sexual Risk Behavior for HIV-Infection
Keywords: HIV-prevention; Internet Prevention intervention; Online randomized controlled trial; Effect evaluation; MSM; Steady relationships

INTERVENTIONS:
Behavioral: Cognitive-behavioral tailored intervention

SUMMARY:
The purpose of this study is to examine the efficacy of a theory based, online tailored intervention on stimulating safe-sex practices among men who have sex with men (MSM). Our hypothesis was that a tailored internet intervention would be more effective in stimulating safe-sex practices of gay men than a non-tailored internet intervention when compared to a waiting-list control group.

DETAILED DESCRIPTION:
Relationships are a high-risk setting for HIV-infection. This trial aimed at testing the efficacy of an online theory-based tailored intervention for preparing single MSM to practice safe sex with future steady partners-labeling it the 'cognitive vaccine approach'.

The target was the promotion of negotiated safety (NS): steady partners testing for HIV and reaching agreements to either be monogamous or to only have safe sex outside the relationship in order to have safe unprotected anal intercourse with each other. The intervention content was based on the information, motivation, behavioral-skills model and the intervention was tailored according to knowledge, motivation, and skill-related deficiencies of each participant. Condom use was promoted as the default alternative for NS. Using an online randomized controlled trial we examined the effects of a tailored versus non-tailored version of the intervention. The cognitive effect (i.e. response efficacy, intentions, and perceived behavioral control (PBC) was measured directly after the intervention and, after 6-months, the behavioral effect (i.e. NS and condom use) via e-mail follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men of all ages, HIV-negative or of unknown serostatus, single, and open to a steady relationship with a man in the future

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 642
Dates: Start 2003-01; Study Completion 2003-08

PRIMARY OUTCOMES:
Scores on the practice of safe sex with steady partners at a six-months follow-up

SECONDARY OUTCOMES:
Scores on response efficacy, intentions and perceived behavioral control regarding the practice of safe sex with steady partners directly after the administration of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Udi Davidovich, Dr., Principal Investigator — Public Health Service of Amsterdam
Locations (1):
- GGD Amsterdam- Amsterdam Health Services, Amsterdam, Netherlands